CLINICAL TRIAL: NCT02272335
Title: Facilitating Adjustment in Low Income Black Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Suzanne C Lechner, Research Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20081005; R01CA131451 (NIH)
Record Dates: First submitted 2014-10-06; First posted 2014-10-22 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Health Disparities; Psychosocial Intervention; Cancer Survivors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CB Stress Management (Experimental): The Cognitive-Behavioral Stress Management (CBSM) intervention arm is a closed, structured group intervention that offers 10 consecutive weekly sessions (and consists of a roughly 30-minute relaxation component, 45-minute cognitive-behavioral stress management component, and a 15-minute break). Groups include an average of 4-9 women and a female African American interventionist. Participants in CBSM receive a workbook that summarizes the rationale for each module, techniques learned within each module, a short out-of-session exercise to practice and the content of the Cancer Wellness and Education (CW) condition as well. i.e. Group Sessions
  Interventions: Behavioral: Group Sessions
- Cancer Wellness (CW) (Active Comparator): Enhanced Breast Cancer Wellness and Education (CW). The CW condition consists of 10 weekly sessions that are roughly 90 minutes in duration. Each session focuses on an important aspect of recovery from breast cancer. Modules were derived from products in the public domain (e.g., National Cancer Institute, Susan G. Komen Foundation, American Cancer Society).i.e. Group Sessions
  Interventions: Behavioral: Group Sessions

INTERVENTIONS:
Behavioral: Group Sessions — 10 weekly sessions:
  * CBSM - 10 consecutive weekly sessions (and consists of a roughly 30-minute relaxation component, 45-minute cognitive-behavioral stress management component, and a 15-minute break). Groups include an average of 4-9 women and a female African American interventionist. Participants in CBSM receive a workbook that summarizes the rationale for each module, techniques learned within each module, a short out-of-session exercise to practice and the content of the CW condition as well.
  * CW/EE - roughly 90 minutes in duration. Each session focuses on an important aspect of recovery from breast cancer. Modules were derived from products in the public domain
  Other Names: CB Stress Management; CW Cancer Wellness

SUMMARY:
The main goal of the proposed study is to test whether a successful stress management intervention can be effectively implemented in natural settings in the community and will be acceptable to a community dwelling, low income population of African American women with breast cancer.

Hypothesis 1: There will be no differences between women randomized to either the Cognitive Behavioral Stress Management (CBSM) or the Cancer Wellness and Education condition (CW) on ratings of acceptability of the program.

Hypothesis 2: Women randomized to the CBSM condition will show greater decreases over time in cancer-specific distress and greater increases over time in quality of life as compared to women in the CW condition over the course of the study from baseline to six month follow-up.

Hypothesis 3: Women randomized to the CBSM condition will show greater improvement in pain levels, sleep disturbance and fatigue as compared to women in the CW condition over the course of the study from baseline to six month follow-up.

Hypothesis 4: Women randomized to the CBSM condition will report fewer sick days, earlier return to work, fewer unanticipated health care visits, fewer visits to the Emergency Department and better follow-up with oncologists as compared to women in the CW condition over the course of the study from baseline to six month follow-up.

Hypothesis 5: Women randomized to the CBSM condition will show more normalized patterns of diurnal cortisol (e.g., greater increase in negative AM-PM slope) as compared to women in the CW condition over the course of the study from baseline to six month follow-up.

Hypothesis 6: Women randomized to the CBSM condition will show more less normalized patterns of heart rate variability (e.g., more variation) as compared to women in the CW condition over the course of the study from baseline to six month follow-up.

DETAILED DESCRIPTION:
Minority women are grossly underserved and suffer poorer quality of life during and after treatment for breast cancer. Despite this greater need, interventions designed to foster adaptation to disease among such women are scarce. Our recent randomized trial tested the efficacy of a 10-week multi-modal, group-based, cognitive behavioral stress management (CBSM) intervention delivered in a university setting among women with breast cancer who recently completed adjuvant treatment. Using a panel of psychological, physiological, and physical indicators of adaptation, the investigators examined whether the intervention facilitated "recovery" or adaptation after adjuvant therapy for breast cancer had been completed. CBSM intervention participants showed improvements in multiple indicators of psychosocial adaptation (fewer intrusive thoughts, lower anxiety, less social disruption, less negative affect, more positive affect, greater benefit finding, and higher levels of positive states of mind), physiological adaptation (decreased cortisol and increased cellular immune function and Th1 cytokine production) and physical adaptation to disease (less fatigue and improved sleep quality). Many of these findings held at 3 and 9 month follow-ups. As with most psychosocial oncology research, participants in the randomized trial were mostly non-Hispanic White women. Whether or not the results of that trial are generalizable to the larger population that includes minority women needs to be tested.

The proposed research aims to translate this University-based, CBSM intervention into a format that will be acceptable and effective in a community setting. The investigators will target our efforts toward low-income African American women, (n=120 after attrition) diagnosed with breast cancer (all stages of disease). Participants will be randomized to 10-week CBSM intervention or an attention time-matched Enhanced Breast Cancer Wellness and Education (CW) active comparison-control condition and monitored for 6 months afterward. Outcomes include: (a) acceptability of the intervention, (b) psychosocial adaptation, (c) physical symptom clusters, (d) economic implications and (e) an objective indicator of stress (diurnal salivary cortisol). The main goal is to test whether a successful stress-management intervention can be effectively implemented in natural settings in the community and will be acceptable to a community-dwelling, low-income population of African American women with breast cancer.

Specific Aim 1: To examine the acceptability of an empirically-validated stress management intervention in community-dwelling low-income African American women with breast cancer.

Specific Aim 2: To test the prediction that participants randomized to CBSM intervention show significant improvements in indices of psychosocial adaptation (i.e., cancer-specific distress, quality of life) relative to women randomized to a CW attention control condition across the study period.

Specific Aim 3: To test the prediction that participants randomized to CBSM intervention show significant improvements in indices of physical symptom clusters relative to women randomized to a CW attention control condition across the study period (physical symptom clusters include pain, sleep, fatigue).

Specific Aim 4: To test the prediction that women randomized to a CBSM intervention versus CW attention control condition have better economic outcomes across the study period (as measured by faster return to work, fewer sick days, fewer health care visits).

Specific Aim 5: To test the prediction that participants randomized to CBSM intervention show significant improvements in indices of physiological adaptation relative to women randomized to a CW attention control condition across the study period by examining diurnal salivary cortisol as objective measure of stress.

ELIGIBILITY:
Inclusion Criteria:

* Women who self-identify as Black;
* No prior history of cancer;
* Age 21 or older;
* Life expectancy of >= 12 months;
* No history of prior inpatient psychiatric treatment for severe mental illness within 1 year (e.g., psychosis)
* No active suicidality;
* No substance dependence within the past year;
* Fluent in English;
* Available for follow-up over the course of the study;
* Endorse moderate stress or distress as measured by a score of 4 or above on the a distress thermometer and an adapted thermometer of stress;
* Completed treatment for breast cancer (except hormonal therapies) within 12 months.

Exclusion Criteria:

* Women who do not self-identify as Black;
* Prior history of cancer (other than skin cancer);
* Under age 21;
* A life expectancy of less than 12 months;
* History of prior inpatient psychiatric treatment for severe mental illness within the past year (e.g., psychosis),
* Active suicidality;
* Substance dependence within the past year;
* Low English fluency;
* Not available for follow-up over the course of the study;
* Score below 4 on a distress thermometer and an adapted thermometer of stress;
* Are not within 12 months of completing treatment for breast cancer (except hormonal therapies) at the time of recruitment;
* Males will be excluded.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Acceptability ratings of the program | 12 months
  Acceptability is measured using a participant self-report scale that was created specifically for this project. This 16-item questionnaire assesses perceived satisfaction with the program, perceived comprehension of the material, comfort with group sessions, perceived competence of the interventionist, satisfaction with project staff, and ratings of project materials on a 4-point Likert scale (completely agree-completely disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C Lechner, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Jackson Health System, Miami, Florida
  - University of Miami, Miami, Florida